CLINICAL TRIAL: NCT00258050
Title: A Four-Way Cross-Over Study to Examine the Effects of Lapatinib on the Pharmacokinetics of Orally and Intravenously Administered Midazolam in Cancer Patients
Brief Title: To Examine The Effects Of Lapatinib On Orally And Intravenously Administered Midazolam In Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EGF10015
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Neoplasms, Breast
Keywords: midazolam; pharmacokinetics; lapatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Midazolam; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with cancer (Experimental): In Part 1 of the study, subjects will be randomized to one of four sequences. All subjects will receive oral or intravenous (IV) midazolam on Days 1, 3, 9 and 11 as per assigned randomization scheme. Starting on Day 4 through Day 11, subjects will receive a daily dose of 1500 milligrams (mg) of oral lapatinib.
  In Part 2, which will begin on Day 12, the subjects will be required to take 1500 mg of lapatinib daily until removed from the study for disease progression, adverse events, withdrawal of consent, or transfer to another lapatinib study.
  Interventions: Drug: Midazolam; Drug: Lapatinib

INTERVENTIONS:
Drug: Midazolam — Subjects will receive midazolam by oral or IV route on Days 1, 3, 9 and 11. Oral midazolam was supplied as 3 mg tablets; IV midazolam was supplied as 1 milligram per milliliter (mg/L) sterile solution.
  Other Names: GW572016 oral tablets
Drug: Lapatinib — Subjects will receive 1500 mg lapatinib by oral route once daily from Day 4.

SUMMARY:
To characterize the effect of repeat oral dose of lapatinib treatment on the pharmacokinetics of a single oral and single intravenous dose of midazolam in adult cancer patients. Also to assess the safety and tolerability of chronic oral lapatinib therapy in cancer patients.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed, solid tumor refractory to standard therapy.
* Tumor for which there is no standard therapy.
* Able to swallow and retain oral medication.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 to 2.
* Provided written informed consent.
* Adequate bone marrow function.
* Serum creatinine is less than or equal to 1.5 mg/dL.
* Calculated creatinine clearance is greater than or equal to 60 ml/min based on Cockcroft and Gault.
* Total bilirubin is greater than or equal to the upper limit of normal of institutional values.
* Aspartate and alanine transaminase is less than or equal to 3 times the upper limit of the institutional values.
* Have a left ventricular ejection fraction (LVEF) greater than or equal to 40% based on electrocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
* Resting oxygen saturations of greater than 90%.

Exclusion criteria:

* Pregnant or lactating female.
* Have malabsorption syndrome, a disease affecting gastrointestinal function.
* Resection of the stomach or small bowel.
* Evidence of symptomatic or uncontrolled brain metastases or leptomeningeal disease.
* Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or screening investigations.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the investigational product.
* Use of anilinoquinazolines, such as gefitinib [Iressa™], erlotinib [Tarceva™].
* Immediate or delayed hypersensitivity reaction to midazolam or any component of the formulation, including benzyl alcohol (cross-sensitivity with other benzodiazepines may exist).
* Has narrow-angle glaucoma which is a contraindication to midazolam use.
* Has received treatment with any investigational drug in the previous 4 weeks.
* Received chemotherapy, immunotherapy, biologic therapy or hormonal therapy within the past 14 days, with the exception of mitomycin C within the past 6 weeks.
* Currently receiving amiodarone or has received amiodarone in the 6 months prior to screening.
* Is taking regular doses of opiates that in the opinion of the investigator would put the patient at risk of clinically significant respiratory compromise when midazolam is administered.
* Physiological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Has Class II to IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Clinically significant electrocardiogram (ECG) abnormality.
* Clinically assessed to have inadequate venous access for protocol-related blood draws.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-11-21 (Actual); Primary Completion 2007-02-08 (Actual); Study Completion 2007-02-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve (AUC) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration. AUC of midazolam in the presence and absence of lapatinib will be determined.
Maximum observed concentration (Cmax) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration. Cmax of midazolam in the presence and absence of lapatinib will be determined.
Clearance (CL) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration. CL of midazolam in the presence and absence of lapatinib will be determined.
Half-life (t½) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration. t1/2 of midazolam in the presence and absence of lapatinib will be determined.
Absolute bioavailability (F) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration. Absolute bioavailability of midazolam in the presence and absence of lapatinib will be determined.

SECONDARY OUTCOMES:
Time of maximum observed concentration (tmax) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration.
Volume of distribution (Vss) of midazolam | Pre-dose, 2 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose on Day 1, Day 3, Day 9 and Day 11
  Blood samples will be collected at indicated time points for the determination of midazolam concentration.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | Up to Month 7
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events may require medical or surgical intervention to prevent one of the other outcomes listed above.
Number of subjects with abnormal clinical chemistry parameters | Up to Month 7
  The following clinical chemistry parameters were evaluated: sodium, potassium, total carbon dioxide (CO2), calcium, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine and blood urea nitrogen (BUN).
Number of subjects with abnormal hematology parameters | Up to Month 7
  The following hematology parameters were evaluated: hemoglobin, hematocrit, red blood cell count, white blood cell count, neutrophil count, lymphocyte count, monocyte count, eosinophil count and basophil count.
Number of subjects with abnormal blood pressure | Up to Month 7
  Systolic and diastolic blood pressure will be measured.
Number of subjects with abnormal heart rate | Up to Month 7
  Heart rate will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Chapel Hill, North Carolina

REFERENCES:
- See also: Results for study EGF10015 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/EGF10015?search=study&search_terms=10015#rs